CLINICAL TRIAL: NCT06948773
Title: A Pilot Study of the Helix Surgical System in Subjects With Primary Open-Angle Glaucoma (POAG) and Cataract.
Brief Title: A Study of the Helix Surgical System in Primary Open-Angle Glaucoma (POAG) and Cataract (HELIX)
Acronym: HELIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09637
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Primary Open Angle Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-arm, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POAG and Cataracts (Experimental): Subjects diagnosed with mild to moderate primary open angle glaucoma (POAG) and cataracts in the study eye.
  Interventions: Device: Helix Surgical System

INTERVENTIONS:
Device: Helix Surgical System — A handheld device to viscodilate up to 360 degrees of Schlemm's canal and collector channels that also enables intracanalicular scaffolding procedure to restore the aqueous outflow system of a glaucomatous eye.

SUMMARY:
A study to assess the safety of the Helix Surgical System in cataract surgery and to gain early evidence of its effectiveness in lowering intraocular pressure (IOP) in subjects with mild to moderate primary open-angle glaucoma (POAG) and cataracts.

DETAILED DESCRIPTION:
To assess the safety of the Helix Surgical System with cataract surgery and gain early evidence on intraocular pressure (IOP) -lowering effectiveness in subjects with mild-moderate primary open-angle glaucoma (POAG) and cataract.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 45 years or older
* Visually significant age-related cataract.
* Intraocular pressure (IOP) at the Screening visit not exceeding 33 mmHg and at least 21 mmHg for unmedicated eyes or 16 mmHg if medicated (1 to 4 ocular hypotensive medications - fixed combinations count as the number of components), with a stable medication regimen for ≥2 months.
* Diagnosed with mild to moderate primary open angle glaucoma (POAG).

Exclusion Criteria:

* Any of the following prior ocular procedures:

  * Laser trabeculoplasty ≤180 days prior to baseline
  * Durysta ≤12 months prior to baseline
  * Any implanted glaucoma device
  * Prior canaloplasty, goniotomy, trabeculotomy, trabeculectomy
  * Ciliary ablation including endoscopic cyclophotocoagulation (ECP), Cyclophotocoagulation or CPC (G probe), high intensity focused ultrasound (HIFU),

    * 180 days prior to baseline
  * Retinal laser procedure ≤3 months prior to baseline
* Any form of glaucoma other than POAG
* Use of topical ocular steroids.
* Clinically significant concurrent ocular pathology or systemic medical condition which, in the Investigator's judgment, would either place the subject at increased risk of complications, contraindicate surgery, place the subject at risk of significant vision loss during the study period or interfere with compliance to elements of the study protocol
* History of penetrating keratoplasty or another corneal transplant
* Endothelial cell density < 2200 cells/mm2 (age 45), < 2000 cells/mm2 (age 46 to 55), < 1800 cells/mm2 (age 56 to 65), < 1600 cells/mm2 (age > 65).
* Retrobulbar tumor, thyroid eye disease, Sturge-Weber Syndrome or any other type of condition that may cause elevated episcleral venous pressure.
* BCVA of logMAR 0.4 (20/50) or worse in the study eye not due to cataract
* BCVA of logMAR 0.6 (20/80) or worse in the non-study eye not due to cataract.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
≥ 20% change from baseline in mean IOP at the 3-month post-operative endpoint | 3 months
  Proportion of subjects with a ≥ 20% change from baseline in mean IOP at the 3-month post-operative endpoint and on the same or fewer medications as preoperatively.

SECONDARY OUTCOMES:
Change in mean IOP | 3 months
  Change in mean IOP at 3 months post-operatively
Average number of ocular hypotensive medications | 3 months
  Average number of ocular hypotensive medications used at 3 months

OTHER OUTCOMES:
Rate of ocular adverse events (AE) | 3 months
  Rate of intraoperative and postoperative ocular adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Dickerson, PhD, Study Director — Sight Sciences, Inc.
Locations (1):
- Panama Eye Center, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No